CLINICAL TRIAL: NCT03074175
Title: Plasma miRNAs Predict Radiosensitivity of Different Fractionation Regimes in Palliative Radiotherapy for Advanced Non-small Cell Lung Cancer：Multicenter Controlled Study.
Brief Title: Plasma miRNAs Predict Radiosensitivity of Different Fractionation Regimes in Palliative Radiotherapy for Advanced Non-small Cell Lung Cancer：Multicenter Controlled Study.(RadmiR-01)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinqiao Hospital of Chongqing (Other)
Responsible Party: Principal Investigator, Jianguo Sun, Deputy director, Xinqiao Hospital of Chongqing
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XQonc-005
Record Dates: First submitted 2017-03-02; First posted 2017-03-08 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Advanced Nsclc
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyperfractionated radiotherapy group (Experimental): According to the size of lung lesions,we divided the patients with lesion ≤5cm in diameterand into hyperfractionated radiotherapy group（50Gy/11F/2W).
  Interventions: Radiation: radiotherapy
- conventional fractionated radiotherapy group (Experimental): According to the size of lung lesions,we divided the patients with lesion >5cm in diameterand into conventional fractionated radiotherapy group（60Gy/30F/6W）.
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — The patient in supine position with hands catch the plate column by crossing the head, and body fixed by vacuum mould. An enhanced 4DCT scan is conducted with a layer thickness and a distance each of 5 mm. the imaging information is input into the Eclipse program system,the gross tumor volume of the primary tumor (GTVt) and pathological lymph nodes (GTVn) are delineated,GTV is expanded in all 3D direction to create PGTV by 5mm margin for squamous cell carcinoma, or an 8mm margin for adenocarcinoma.Radiaion therapy is delivered by 5F-IMRT.For conventional fractionated radiotherapy,the prescribed dose covering 95% of PGTV is 60Gy/30F/6W.For hyperfractionated radiotherapy,the prescribed dose covering 95% of PGTV is 50Gy/11F/2W.lung V20 <25%, lung V30 <18%, spinal cord <36 Gy.

SUMMARY:
Lung cancer is a malignant tumor that causes the highest morbidity and mortality, and the main pathological type is non-small cell lung cancer (NSCLC). Most of them present with advanced stage at diagnosis. Radiotherapy is an important treatment strategy for advanced non-small cell lung cancer. However patients have different responses to radiotherapy due to individual differences, thus there is still lacking of sensitive markers to predict treatment response at present. Using bioinformatics to process the data and small sample clinical trial, our previous study found 5 plasma miRNAs were related to radiosensitivity. The design is controlled clinical trial. According to the size of lung lesions, the investigators divided the patients into hyperfractionated radiotherapy group（50Gy/11F/2W) with lesion ≤5cm in diameter and conventional fractionated radiotherapy group（60Gy/30F/6W）with lesion >5cm in diameter.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological histology and/or cytology confirmed NSCLC;
2. Based on AJCC Cancer Staging, IIIA, IIIB, IV lung cancer patients with NSCLC;
3. PS 0-2;
4. Expected survival > 3 months;
5. Age 18~75 years old;
6. The function of lung, liver, kidney, bone marrow was normal;
7. The patients had not received radiotherapy for previous primary tumor and metastases;
8. At least accept 2-4 cycles of chemotherapy,not disease progression after chemotherapy,start radiotherapy in two weeks after the last cycle of chemotherapy;
9. Wild-type EGFR;
10. Sensitive mutant EGFR, but refused to targeted therapy;
11. In line with the indications of radiotherapy and accept it;
12. Voluntarily enrolled to participate in,better compliance, cooperate with experimental observations, and sign informed consent.

Exclusion Criteria:

1. Vital organs (e.g., heart, liver, kidney) have serious dysfunction;
2. Patients with other malignancies;
3. Patients with a history of autoimmune disease;
4. The patients are pregnant and lactating (Women of childbearing age need to check the pregnancy test);
5. In the activity of acute or chronic infectious diseases;
6. Patients with a clear history of drug allergy or allergic genus;
7. Patients with participating in other clinical trials at the same time;
8. Other cases that researchers believe that patients should not participate in the present trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | up to two and a half years

SECONDARY OUTCOMES:
Correlation between the expression level of miRNAs and the ORR. | up to two and a half years
Progression free survival（PFS） | up to two and a half years
side effects of radiation | up to two and a half years

CONTACTS AND LOCATIONS:
Locations (1):
- Xinqiao Hospital of Chongqing, Chongqing, China